CLINICAL TRIAL: NCT01954862
Title: Comparison of Methods for Luminal Distention for on Demand Sedation Colonoscopy: Air Insufflation, Carbon Dioxide and Water-aided Colonoscopy. A Randomized Controlled Trial.
Brief Title: Comparison of Methods to Distend the Colon During Insertion: CO2, Air Insufflation, Water-aided Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Presidio Ospedaliero Santa Barbara (Other)
Responsible Party: Principal Investigator, Sergio Cadoni, M.D., Responsabile Servizio Endoscopia Digestiva, Presidio Ospedaliero Santa Barbara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG. 2013/3403
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Pain; Colorectal Adenomas; Colorectal Cancer
Keywords: Water-aided colonoscopy; Water Immersion colonoscopy; Water Exchange colonoscopy; Carbon-dioxide colonoscopy; Painless unsedated colonoscopy; Adenoma detection rate; Mean Adenomas per Procedure
MeSH Terms: conditions — Pain; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Air insufflation method. (Active Comparator): Colonoscopy performed in the standard fashion, with the minimal air insufflation required to aid insertion and allowing for washing as needed. Considered to be standard procedure.
  Interventions: Other: Air Insufflation method.
- CO2 insufflation (Experimental): Colonoscopy performed with CO2 insufflation using the insufflation unit, allowing for washing as needed.
  Interventions: Other: CO2 insufflation
- Water Immersion/CO2 (Experimental): Infusion of water during the insertion phase of colonoscopy mainly to open the colonic lumen and progress to the cecum immersed in the water environment thus created, without attempting to clear the colon contents. Residual air in the colon will not be removed. Infused water and residual feces will be suctioned back predominantly during withdrawal. Insufflation not used until the cecum is reached. It will be allowed only 3 times and no more than 10 seconds each time (ITT failure if >3) if the lumen cannot be seen. Withdrawal phase done using CO2 insufflation.
  Interventions: Other: Water Immersion/CO2
- Water Exchange/CO2 (Experimental): Insufflation not used until the cecum is reached. Infusion of a sufficient amount of water to render the lumen of the colon a slit to progress with the colonoscope. Part of the infused water will be constantly suctioned back exchanging clean for dirty or hazy water. Air pockets will be always aspirated to collapse the lumen. After cecal intubation as much residual water as possible will be aspirated before beginning the withdrawal phase. During withdrawal residual water and feces will be suctioned. Withdrawal phase done using CO2 insufflation.
  Interventions: Other: Water Exchange/CO2
- Water Immersion/AI (Experimental): Infusion of water during the insertion phase of colonoscopy mainly to open the colonic lumen and progress to the cecum immersed in the water environment thus created, without attempting to clear the colon contents. Residual air in the colon will not be removed. Infused water and residual feces will be suctioned back predominantly during withdrawal. Insufflation not used until the cecum is reached. It will be allowed only 3 times and no more than 10 seconds each time (ITT failure if >3) if the lumen cannot be seen. Withdrawal phase done using room air insufflation.
  Interventions: Other: Water Immersion/AI
- Water Exchange/AI (Experimental): Insufflation not used until the cecum is reached. Infusion of a sufficient amount of water to render the lumen of the colon a slit to progress with the colonoscope. Part of the infused water will be constantly suctioned back exchanging clean for dirty or hazy water. Air pockets will be always aspirated to collapse the lumen. After cecal intubation as much residual water as possible will be aspirated before beginning the withdrawal phase. During withdrawal residual water and feces will be suctioned. Withdrawal phase done using room air insufflation.
  Interventions: Other: Water Exchange/AI

INTERVENTIONS:
Other: Air Insufflation method. — Air Insufflation method.
  Arms: Air insufflation method.
Other: CO2 insufflation — CO2 insufflation.
  Arms: CO2 insufflation
Other: Water Immersion/CO2 — Water Immersion during insertion, CO2 insufflation during withdrawal.
  Arms: Water Immersion/CO2
Other: Water Exchange/CO2 — Water Exchange during insertion, CO2 insufflation during withdrawal.
  Arms: Water Exchange/CO2
Other: Water Immersion/AI — Water Immersion during insertion, AI insufflation during withdrawal.
  Arms: Water Immersion/AI
Other: Water Exchange/AI — Water Exchange during insertion, AI insufflation during withdrawal.
  Arms: Water Exchange/AI

SUMMARY:
Insufflation of the colon, usually with room air, is necessary to distend the lumen for exploration. Carbon dioxide (CO2) insufflation instead of room air insufflation (AI) has been shown to decrease symptoms of abdominal pain or discomfort during the procedure and particularly during the following 24 hours. CO2 is is rapidly absorbed by the intestinal mucosa and exhaled through respiration. AI colonoscopy has usually been the reference standard to compare colonoscopy using CO2 insufflation. In two recent articles AI was compared to either CO2 insufflation and Water-aided colonoscopy (WAC), which entails infusion of water to facilitate insertion to the cecum.

WAC can be categorized broadly in Water Immersion (WI) and Water Exchange (WE). In WI water is infused during the insertion phase of colonoscopy, with removal of infused water predominantly during withdrawal. Occasional use of insufflation may be allowed. WE entails complete exclusion of insufflation, removal of residual colonic air pockets and feces, and suction of infused water predominantly during insertion to minimize distention. During the withdrawal phase insufflation is used to distend the colonic lumen.

In the WAC arms of the two mentioned articles the insertion method used was WI, with infusion of water at room temperature or at 37°C. During withdrawal, air insufflation or either air or CO2 insufflation were employed.

Compared to AI, CO2 insufflation and WI (using room air insufflation or CO2 insufflation during withdrawal) were effective in both studies in decreasing sedation requirement, pain and tolerance scores, with patients' higher willingness to repeat the procedure.

Until now no direct comparison has been made within a single study about pain score during colonoscopy using AI, CO2 insufflation, WI/CO2, WE/CO2, WI/AI and WE/AI.

In this study we test the hypothesis that, compared to AI, CO2 insufflation and WAC/CO2-AI methods will decrease pain score during colonoscopy, with reduction of sedation requirement, and that WE will achieve the best result. This comparative study has also the aim to test the respective peculiarities of each method.

DETAILED DESCRIPTION:
Design: Prospective double blinded two-center randomized controlled trial. Methods: Colonoscopy with air insufflation, CO2, Water Immersion/CO2, Water Exchange/CO2, Water Immersion/AI and Water Exchange/AI to aid insertion of colonoscope; split dose bowel preparation; on demand-sedation.

Control method: Air insufflation colonoscopy. Study methods: CO2 colonoscopy, Water Immersion/CO2 colonoscopy, Water Exchange/CO2 colonoscopy, Water Immersion/AI colonoscopy, Water Exchange/AI colonoscopy.

Population: Consecutive 18 to 85 year-old diagnostic in-patients and outpatients. After informed consent, assignment to control or study arms based on computer generated randomization list with block allocation and stratification.

Primary outcome: Maximum pain score recorded during colonoscopy. Secondary outcomes: Cecal intubation rate and time, total procedure time (including biopsy and/or polypectomy), need for sedation and its dosage, overall pain score at discharge. In addition, Adenoma Detection Rate, Mean Adenomas per Procedure, position changes, amount of infused and suctioned water during insertion and withdrawal will be recorded. Bloating after examination and at discharge and patient willingness to repeat the examination will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive 18 to 85 year-old diagnostic in-patients and outpatients agreeing to start procedure without premedication.

Exclusion Criteria:

* Patient unwillingness to start the procedure without sedation/analgesia
* previous colorectal surgery
* proctosigmoidoscopy or bidirectional endoscopy
* patient refusal or inability to provide informed consent
* inadequate assumption of bowel preparation
* moderate or severe chronic obstructive pulmonary disease requiring oxygen
* medical history of CO2 retention

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Maximum pain score recorded during colonoscopy. | 1 hour
  Pain assessed using a visual analogue scale (VAS) with a score 0=absence of pain, 2=simply "discomfort", 10=the worst possible pain. Before the procedure, an endoscopic nurse will explain the VAS scoring system to the patients. Every 60 seconds during colonoscopy patients will be asked about discomfort or pain. The responses will be recorded, and the maximum pain score noted.

SECONDARY OUTCOMES:
Overall pain after the procedure. | 1 hour.
  After the procedure and at discharge from the Endoscopy Unit, an assistant nurse blinded to the procedure will ask patients about overall pain using the same VAS when neither the endoscopist nor the assistant nurse who performed the colonoscopy will be present. Patients will be asked to quantify the degree of pain experienced and to place a mark over the VAS accordingly.
Cecal intubation rate. | 1 hour
  Cecal intubation will be defined as passage of the tip of the colonoscope beyond the ileocecal valve so that the medial wall of the cecum proximal to the ileocecal valve will be observed.
Cecal intubation time. | 1 hour.
  Cecal intubation time will be defined as the time for passage of the colonoscope from the rectum to the cecum.
Total procedure time. | 1 hour.
  Total procedure time (including time required for polyp resection or biopsy).
Adenoma detection rate. | 15 months.
  Proportion of subjects with at least one adenoma of any size.
Mean adenomas per procedure. | 15 months.
  Total number of adenomas resected per subject.
Advanced adenomas. | 15 months.
  Total number of advanced adenomas: diameter ≥10mm, or high grade dysplasia, or with ≥20% villous components.

OTHER OUTCOMES:
Position changes. | 1 hour.
  Change in patient position as needed if advancement of the colonoscope fails.
Loop reduction maneuvers. | 1 hour.
  Applied as needed if advancement of the colonoscope fails.
Amount of water used during the procedure. | 1 hour.
  Amount of water infused and aspirated during insertion and withdrawal.
Bloating at completion of examination. | 1 hour.
  Bloating felt by patients at completion of examination on a 10 point visual analogue scale.
Bloating at discharge. | 1 hour.
  Bloating felt by patients at discharge measured on a ten point visual analogue scale.
Patients willingness to repeat the examination. | 1 hour.
  Patients willingness to repeat the examination based on overall satisfaction about procedure. Measured at discharge on a yes/no question.
Oxygen desaturation. | 1 hour.
  Significant oxygen desaturation will be recorded when values less than 85% will be maintained for more than 15 seconds.
Vagal reaction. | 1 hour.
  Vagal reaction is defined as heart rate <60 beats per minute accompanied by excessive sweating, nausea and/or vomiting.
Abdominal Compression. | 1 hour.
  Compression of abdomen if advancement of the colonoscope fails.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Cadoni, MD, Principal Investigator — S. Barbara Hospital, Iglesias (CI), Italy
Locations (3):
- Sepulveda Ambulatory Care Center, VA Greater Los Angeles Healthcare System, Los Angeles, California, United States
- Vìtkovice Hospital, Ostrava, Czechia
- S. Barbara Hospital, Iglesias, CI, Italy

REFERENCES:
- [Background] Falt P, Liberda M, Smajstrla V, Kliment M, Bartkova A, Tvrdik J, Fojtik P, Urban O. Combination of water immersion and carbon dioxide insufflation for minimal sedation colonoscopy: a prospective, randomized, single-center trial. Eur J Gastroenterol Hepatol. 2012 Aug;24(8):971-7. doi: 10.1097/MEG.0b013e3283543f16. PMID 22569079
- [Background] Amato A, Radaelli F, Paggi S, Baccarin A, Spinzi G, Terruzzi V. Carbon dioxide insufflation or warm-water infusion versus standard air insufflation for unsedated colonoscopy: a randomized controlled trial. Dis Colon Rectum. 2013 Apr;56(4):511-8. doi: 10.1097/DCR.0b013e318279addd. PMID 23478620
- [Background] Leung FW, Amato A, Ell C, Friedland S, Harker JO, Hsieh YH, Leung JW, Mann SK, Paggi S, Pohl J, Radaelli F, Ramirez FC, Siao-Salera R, Terruzzi V. Water-aided colonoscopy: a systematic review. Gastrointest Endosc. 2012 Sep;76(3):657-66. doi: 10.1016/j.gie.2012.04.467. PMID 22898423
- [Background] Rabenstein T, Radaelli F, Zolk O. Warm water infusion colonoscopy: a review and meta-analysis. Endoscopy. 2012 Oct;44(10):940-51. doi: 10.1055/s-0032-1310157. Epub 2012 Sep 17. PMID 22987214
- [Background] Leung FW. Water-aided colonoscopy. Gastroenterol Clin North Am. 2013 Sep;42(3):507-19. doi: 10.1016/j.gtc.2013.05.006. PMID 23931857
- [Background] Wu J, Hu B. The role of carbon dioxide insufflation in colonoscopy: a systematic review and meta-analysis. Endoscopy. 2012 Feb;44(2):128-36. doi: 10.1055/s-0031-1291487. Epub 2012 Jan 23. PMID 22271023
- [Background] Dellon ES, Hawk JS, Grimm IS, Shaheen NJ. The use of carbon dioxide for insufflation during GI endoscopy: a systematic review. Gastrointest Endosc. 2009 Apr;69(4):843-9. doi: 10.1016/j.gie.2008.05.067. Epub 2009 Jan 18. PMID 19152906
- [Derived] Cadoni S, Falt P, Gallittu P, Liggi M, Mura D, Smajstrla V, Erriu M, Leung FW. Water Exchange Is the Least Painful Colonoscope Insertion Technique and Increases Completion of Unsedated Colonoscopy. Clin Gastroenterol Hepatol. 2015 Nov;13(11):1972-80.e1-3. doi: 10.1016/j.cgh.2015.04.178. Epub 2015 May 5. PMID 25956838